CLINICAL TRIAL: NCT01400646
Title: An Open-Label, Non-Randomized, Sequential Two-Treatment Period Study to Explore the Pharmacodynamic Changes When Transitioning From Rivaroxaban to Warfarin
Brief Title: A Study to Explore the Pharmacodynamic Changes When Transitioning From Rivaroxaban to Warfarin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR018664; RIVAROXAFL1004 (Other: Janssen Research & Development); 2011-002890-46 (EudraCT Number); NCT01510925 (obsolete NCT alias)
Record Dates: First submitted 2011-07-21; First posted 2011-07-22 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Healthy
Keywords: Rivaroxaban; JNJ-39039039; BAY59-7939; Warfarin; Transition
MeSH Terms: interventions — Rivaroxaban; Warfarin; Vitamin K

ARMS (2):
- Rivaroxaban + Warfarin Concomitant Therapy Phase (Experimental): Rivaroxaban monotherapy 20 mg/day for 5 days followed by Rivaroxaban 20 mg/day + Warfarin. 10 mg/day for >= 2 to <= 4 days concomitant therapy, then Warfarin monotherapy 0-15 mg/day for 4 days (Treatment Period 1). A 14-day washout period will separate Treatment Periods 1 and 2.
  Interventions: Drug: Rivaroxaban; Drug: Warfarin; Drug: Vitamin K
- Warfarin Monotherapy Phase (Experimental): Warfarin monotherapy 10 mg/day for >=2 to <=4 days, then Warfarin 0-15 mg/day for 4 days (Treatment Period 2). A 14-day washout period will separate Treatment Periods 1 and 2.
  Interventions: Drug: Vitamin K; Drug: Warfarin

INTERVENTIONS:
Drug: Rivaroxaban — Type=exact number, unit=mg, number=20, form=tablet, route=oral use. One tablet once daily for 5 days (Treatment Period 1, Days 1-7).
  Arms: Rivaroxaban + Warfarin Concomitant Therapy Phase
Drug: Warfarin — Type=exact number, unit mg, number=10, form=tablet , route=oral use. One tablet for 2-4 days (Treatment Period 1, Day 6 up to Day 11).
  Arms: Rivaroxaban + Warfarin Concomitant Therapy Phase
Drug: Vitamin K — Type=exact number, unit=mg, number=1, form=oral solution, route=oral use. 1 mg dose for 1 day (Treatment Period 1, Day 12).
  Arms: Rivaroxaban + Warfarin Concomitant Therapy Phase
Drug: Vitamin K — Type=exact number, unit=mg, number=5, form=oral solution, route=oral use. 5 mg dose for 1 day (Treatment Period 2, Day 7).
  Arms: Warfarin Monotherapy Phase
Drug: Warfarin — Type-exact number, unit=mg, number=10, form=tablet, route=oral use. Tablet(s) administered once daily for 2-4 days (Treatment Period 2, Day 1 up to Day 6)
  Arms: Warfarin Monotherapy Phase
Drug: Warfarin — Type=range, unit=mg, number=0-15, form=tablet, route=oral use. Tablet(s) taken once daily for up to 4 days after Warfarin 10 mg administered as monotherapy for 2-4 days (Treatment Period 1).
  Arms: Rivaroxaban + Warfarin Concomitant Therapy Phase
Drug: Warfarin — Type=range, unit=mg, number=0-15, form=tablet, route=oral use. Tablet(s) taken once daily for up to 4 days after Warfarin 10 mg administered as monotherapy for 2-4 days (Treatment Period 2).
  Arms: Warfarin Monotherapy Phase

SUMMARY:
The purpose of this study is to explore the pharmacodynamic (what the drug does to the body) changes when transitioning from rivaroxaban 20 mg once daily to warfarin dosed to a therapeutic level as measured by the International Normalized Ratio (INR) range of 2.0 to 3.0 in healthy volunteers. In addition, the pharmacokinetics (what the body does to the drug), safety and tolerability of rivaroxaban during the transition to warfarin will be investigated. The INR is obtained from a blood test, and is a measure for the clotting tendency of the blood used for safe and adequate dosing of warfarin.

DETAILED DESCRIPTION:
This is a single-center, open-label (study staff and healthy volunteers will know the identity of treatment assigned), sequential 2-treatment period study in healthy adult volunteers to explore the pharmacodynamic changes (changes drugs have on the body), specifically in regard to blood coagulation (blood clotting) when healthy volunteers take oral (by mouth) rivaroxaban followed by warfarin. Treatment Period 1: Rivaroxaban 20 mg/day for 5 days then Rivaoxaban 20 mg/day + Warfarin 10 mg/day for 2-4 days then warfarin 0-15 mg/day for 4 days. Treatment Period 2: Warfarin 10 mg/day for 2-4 days, then 0-15 mg/day for 4 days. Treatment periods 1 and 2 will be separated by a washout period of at least 14 days. In Treatment Periods 1 and 2, the dose of warfarin may be adjusted as specified by the protocol and the last dose of warfarin in each Treatment period will be followed by a single dose of Vitamin K. The approximate total study length for healthy adult volunteers enrolled is approximately 72 days (includes a 28-day Screening Period, a 30-day Open-label Treatment Phase, which includes the 7 days for a follow-up visit, and at least a 14-day washout between treatment periods).

ELIGIBILITY:
Inclusion Criteria:

* Volunteers must agree to provide a blood sample for pharmacogenomic testing and must have less than 3 of the variant CYP2C9 and VKORC1 gene alleles associated with increased warfarin sensitivity if their genetic status regarding these alleles is not previously known
* Have coagulation test results (INR, PT, and activated partial thromboplastin time (aPTT) within clinically acceptable limits, blood pressure (after the volunteer is supine for 5 minutes) between 90 and 140 mmHg systolic, inclusive, and between 50 and 90 mmHg diastolic
* Have a body mass index (BMI) between 18 and 30 kg/m2 (inclusive), and body weight of not less than 50 kg
* Be a Non-smoker (Volunteers may not use nicotine-containing products within 3 months prior to study drug administration

Exclusion Criteria:

* Have a history or current clinically significant medical illness, including (but not limited to) of intracranial tumor or aneurysm
* Have history of gastrointestinal disease (e.g., Crohn's disease) which could result in impaired absorption of the study drugs or history of clinically significant hemoptysis, excessive bruising, bleeding from nose or gums or known disorders with increased bleeding risk (e.g., acute gastritis, acute peptic ulcer) or history of any bleeding diathesis. Concomitant use (also within the last 2 weeks before start of the study) of drugs that influenced the coagulation system, e.g., antiplatelet drugs (e.g., acetylsalicylic acid, ticlopidine and clopidogrel
* abciximab, tirofiban and integrelin) or other anticoagulants (antithrombins, unfractionated heparins, low molecular weight heparins and hirudin, coumadin-type anticoagulants phenprocoumon, warfarin, dabigatran, probenecide)
* Use of medications known to affect the metabolic pathways (CYP3A4, or P-gp) within 14 days of study admission

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2011-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Prothrombin time (PT) | From Day 1 up to Day 9
International Ratio (INR) | From Day 1 up to Day 9

SECONDARY OUTCOMES:
Plasma concentrations of Rivaroxaban | Up to Day 9
Plasma concentrations of Warfarin | Up to Day 12

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium

REFERENCES:
- [Derived] Moore KT, Byra W, Vaidyanathan S, Natarajan J, Ariyawansa J, Salih H, Turner KC. Switching from rivaroxaban to warfarin: an open label pharmacodynamic study in healthy subjects. Br J Clin Pharmacol. 2015 Jun;79(6):907-17. doi: 10.1111/bcp.12559. PMID 25475601